CLINICAL TRIAL: NCT00357617
Title: Evaluation of the Effect of Celecoxib on Angiogenesis Markers in Patients With Operable Head and Neck Squamous Cell Carcinoma
Brief Title: Celecoxib in Treating Patients With Head and Neck Cancer That Can Be Removed By Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000490047; CHUV-CEPO-161-05; EU-20627
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2008-01

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Celecoxib; Microarray Analysis; Immunoenzyme Techniques; Immunohistochemistry; Biopsy; Neoadjuvant Therapy

INTERVENTIONS:
Drug: celecoxib
Genetic: microarray analysis
Genetic: protein expression analysis
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving celecoxib before surgery may reduce the amount of normal tissue that needs to be removed. Collecting and storing samples of tumor tissue, blood, and urine from patients with head and neck cancer to study in the laboratory may help doctors learn more about the cancer and predict how well patients will respond to treatment with celecoxib.

PURPOSE: This phase I/II trial is studying changes in tumor cells and how well celecoxib works in treating patients with head and neck cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the changes in molecular markers of angiogenesis before and after treatment with celecoxib in tumor tissues of patients with resectable head and neck squamous cell carcinoma.

Secondary

* Evaluate the changes in molecular markers of angiogenesis before and after treatment with celecoxib in blood tissues of these patients.
* Evaluate the effects of celecoxib on indirect measures of tumor perfusion, as measured by perfusion CT scan, in these patients.
* Evaluate the effects of celecoxib on apoptosis and proliferation rate on tumor cells and on endothelial cells in these patients.
* Identify potential new markers of the activity of cyclooxygenase-2 inhibitors and identify new pathways of potential interests by performing gene expression profiling of tumor tissues before and after exposure to celecoxib.

OUTLINE: This is an open-label, nonrandomized, uncontrolled study.

Patients undergo panendoscopy and tumor biopsy on day 0. Patients receive oral celecoxib twice daily beginning on day 1 and continuing for at least 14 days*. Patients then undergo definitive surgery.

NOTE: *Treatment continues until the day before surgery.

Tumor, blood, and urine samples are collected at baseline and periodically during study. Tumor quantification by perfusion CT scan is performed at baseline and after treatment with celecoxib. Biological markers are detected by immunohistochemistry and enzyme immunoassay. Blood vascular density, apoptosis, proliferation, and endothelial cell:tumor ratio are measured by indirect hemagglutination. Gene expression is measured by microarray analysis.

After surgery, patients are followed at 4 weeks and then periodically thereafter.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed or high clinical suspicion of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx

  * No carcinoma of sinonasal or nasopharynx
* Clinical stage T1-4, N0-2, M0 disease

  * Tumor must be considered resectable with planned surgical excision
  * No lymph nodes > 6 cm (N3)
  * No distant metastasis

PATIENT CHARACTERISTICS:

* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 60 mL/min
* AST and ALT ≤ 2.5 times ULN
* Bilirubin normal
* History of prior malignancy allowed if there is no evidence of recurrence or metastases at the time of screening
* No comorbidity that precludes operability
* No known liver impairment
* Known recent gastric or duodenal ulcer allowed if treated for > 6 weeks prior to study enrollment
* No known hypersensitivity to celecoxib
* No known allergic reactions to sulfonamides, aspirin, or other NSAIDs
* No psychological, familial, sociological, or geographical condition that would interfere with study compliance and follow-up schedule
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* More than 2 months since prior and no other concurrent anticancer or investigational drugs
* More than 2 weeks since prior and no other concurrent nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids
* No prior radiotherapy to the head and neck region
* No concurrent radiotherapy
* No concurrent therapeutic anticoagulation
* No concurrent administration of any of the following:

  * Other cyclooxygenase-2 inhibitors
  * Aspirin

    * Low-dose aspirin for cardiovascular prophylaxis allowed
  * Aluminum and magnesium-containing antacids
  * ACE inhibitors
  * Furosemide
  * Known inhibitors of P450 2C9 (e.g., fluconazole, fluoxetine, fluvoxamin, isoniazid, omeprazole)
  * Known inducers of P450 2C9 (e.g., rifampin)
  * Lithium
  * Acenocoumarol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
Molecular markers of angiogenesis in tumor tissues (PGE2, VEGF, MMP-9, sFlt-1, ERK phosphorylation, PKB phosphorylation, and ErbB2 levels)

SECONDARY OUTCOMES:
Molecular markers in plasma (VEGF, MMP-9, and sFlt1)
Molecular marker in urine (PGE2)
Apoptosis/proliferation in tumor cells and endothelial cells
Gene expression profiling in fresh tumor tissues (Erb-B2, c-IAP-2, PAI-1, MAPK-4, integrin α V, N-CAM, caspase 6, ErbB2 transducer, angiopoietin like-2, interleukin-8, and MMP13)
Tumor perfusion imaging by perfusion CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Francois Luthi, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland